CLINICAL TRIAL: NCT06218433
Title: Urothelial Cancer Screening in Individuals With Lynch Syndrome Using a Urine Tumor DNA Panel (LS-URO Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: R22125; R22125 (Other: Tampere University Hospital)
Record Dates: First submitted 2024-01-10; First posted 2024-01-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Urothelial Carcinoma; Lynch Syndrome
Keywords: Lynch syndrome; Hereditary cancer syndrome; Screening; Urothelial neoplasms; Bladder neoplasms; Upper tract urothelial neoplasms; Urogenital diseases; Liquid biopsies; Urine tumor DNA
MeSH Terms: conditions — Carcinoma, Transitional Cell; Colorectal Neoplasms, Hereditary Nonpolyposis; Neoplastic Syndromes, Hereditary; Urinary Bladder Neoplasms; Urogenital Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening arm (Experimental): Invitation to participate in urothelial cancer screening and questionnaires
  Interventions: Diagnostic Test: Urothelial cancer screening using urine tumor DNA test; Diagnostic Test: Urothelial cancer screening using urine cytology (comparator)

INTERVENTIONS:
Diagnostic Test: Urothelial cancer screening using urine tumor DNA test — Urine sample DNA is analyzed using a targeted sequencing panel encompassing the coding regions of 21 genes that are recurrently mutated in urothelial cancer
Diagnostic Test: Urothelial cancer screening using urine cytology (comparator) — Urine cytology sample

SUMMARY:
Lynch syndrome (LS) is an inherited cancer predisposition syndrome caused by pathogenic germline variants in DNA mismatch repair (MMR) genes. New cancer screening and diagnostic tools are urgently needed to identify LS-related cancers early enough for curative treatment. Urothelial cancers (comprising bladder and upper tract urothelial tumors) are the third most common cancer after colorectal and endometrial cancers in individuals with LS. Up to one in four LS individuals will develop urothelial cancer during their lifetime, with the risk varying based on the defective MMR gene. In this clinical trial, we will employ urine tumor DNA (utDNA) to identify asymptomatic urothelial cancers in Lynch syndrome patients, and to investigate the potential benefits of urine tumor DNA based screening in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Diagnosis of Lynch syndrome
* Age 50 - 75 years at study recruitment

Exclusion Criteria:

* Concurrent urothelial carcinoma

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of positive utDNA for urothelial cancer within one year of follow-up | At 1 years of follow-up
  Sensitivity and specificity of positive utDNA for urothelial cancer, using histologically verified cancers detected within 1 year of the utDNA test as ground truth

SECONDARY OUTCOMES:
Specificity of positive utDNA for urothelial cancer at the time of testing | After all patients with positive utDNA have been evaluated with cystoscopy and/or imaging
  Specificity of positive utDNA test for urothelial cancer, using histologically verified cancers detected in the cystoscopy and/or imaging performed due to positive utDNA test as the ground truth
Sensitivity and specificity of positive utDNA for urothelial cancer within multiple years of follow-up | At 2, 5, and 10 years of follow-up
  Sensitivity and specificity of positive utDNA for urothelial cancer, using histologically verified cancers detected within 2, 5, and 10 years of the utDNA test as ground truth
Overall survival | At 5 and 10 years of follow-up
  Overall survival in utDNA positive and negative patients
Urothelial cancer specific survival | At 3, 5 and 10 years of follow-up
  Urothelial cancer specific survival survival in utDNA positive and negative patients
Time to metastatic urothelial cancer | At 5 and 10 years of follow-up
  Time to metastatic urothelial cancer in utDNA positive and negative patients
Time to diagnosis of muscle invasive or high grade urothelial cancer | At 2, 5 and 10 years of follow-up
  Time to diagnosis of muscle invasive or high grade urothelial cancer in utDNA positive and negative patients
Time to diagnosis of urothelial cancer | At 2, 5 and 10 years of follow-up
  Time to diagnosis of urothelial cancer in utDNA positive and negative patients
TNM pathological stage of urothelial cancers | At 2, 5 and 10 years of follow-up
  TNM pathological stage (American Joint Committee on Cancer (AJCC)/International Union Against Cancer (UICC)) of urothelial cancers found in utDNA positive and negative patients
Size of urothelial tumors | At 2, 5 and 10 years of follow-up
  Maximum diameter of urothelial tumors found in utDNA positive and negative patients
Urothelial cancer grade | At 2, 5 and 10 years of follow-up
  The World Health Organization (WHO) 2004/2016 grading of urothelial cancers found in utDNA positive and negative patients

OTHER OUTCOMES:
Sensitivity and specificity of urine cytology | At 1 year of follow-up
  Sensitivity and specificity of urine cytology for detecting urothelial cancer, using histologically verified cancers detected within 1 year of cytology as ground truth
Association of utDNA fraction with time to diagnosis of urothelial cancer | At 2, 5 and 10 years of follow-up
  Association of utDNA fraction (quantified based on mutation allele fractions in urine DNA) with time to diagnosis of urothelial cancer
Prevalence of somatic second hit in MMR genes | At 1, 2, 5 and 10 years of follow-up
  Prevalence of somatic second hit and additional somatic hits in mismatch repair genes (MSH2, MSH6, MLH1, PMS2) in Lynch syndrome patients diagnosed with urothelial cancer
Cost of utDNA screening | At 1, 2, 5 and 10 years of follow-up
  Analysis of the cost of utDNA screening, including cost per urothelial cancer found

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Nikkola, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (2):
- Vancouver Prostate Centre, Vancouver, Canada
- Tampere University Hospital and Tampere University, Tampere, Finland